CLINICAL TRIAL: NCT00637117
Title: A Phase I/II Study of Intratumoral Dendritic Cell Vaccination Combined With Local Radiotherapy in Patients With Recurrent Lymphoma.
Brief Title: Intratumoral Dendritic Cell Vaccination Combined With Local Radiotherapy in Patients With Recurrent Lymphoma.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study never opened and not sure if it ever will.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Wenru Song, MD, PhD, Baylor Institute for Immunology Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007-082
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Lymphoma
Keywords: Lymphoma, Dendritic, Vaccine, Radiotherapy
MeSH Terms: conditions — Lymphoma | interventions — Interferon-alpha; Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Autologous dendritic cells generated using GM-CSF, interferon alpha and LPS — Day 1 and Day 2: 2 Gy Radiation on Day 1 and Day 2 to tumor site. Day 4, 8, 11, 18: 0.5mL injection of Autologous dendritic cells generated using GM-CSF, interferon alpha and LPS.

SUMMARY:
The purpose of the study is to gather data on feasibility and on immune and clinical efficacy of intratumoral dendritic cell (DC) vaccination in combination with local radiotherapy in patients with recurrent lymphoma

DETAILED DESCRIPTION:
Lymphoma is extremely sensitive to radiation and is a commonly used therapy. The major issue in application of local radiotherapy is the relative short duration of response and as a consequence is used mainly for palliation. Therefore novel therapies are needed to improve the outcome of patients with lymphomas. The potential specificity of the immune system to recognize and eliminate tumor cells is especially relevant in lymphoma. Immune responses are induced, coordinated and regulated by dendritic cells (DCs), the most potent antigen-presenting cells. Based on the central role of DCs in initiating immune responses, four vaccinations will be administered at intervals beginning two days after low dose radiation is given to the tumor site.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed recurrent lymphoma of any initial stage, either Hodgkin's lymphoma or the B cell or T cell NHL of an indolent nature. For B cell lymphoma, follicular lymphoma, small lymphocytic lymphoma, marginal zone lymphoma, and those indolent patients with mantle cell lymphoma or diffuse large B cell lymphoma will be included. For T cell lymphoma, the patients with indolent cutaneous T cell lymphomas (mycosis fungoides or primary cutaneous anaplastic large cell lymphoma) who have failed or have been intolerant of one systemic or two topical treatments will be included.
* Patients must have failed at least one line of prior treatment but not more than four (including autologous but not allogeneic stem cell transplant).
* Patients must have at least one site of disease that is accessible for intratumoral injection of DCs percutaneously after palliative local radiotherapy
* Tumor specimens must be available for immunological studies either from a previous biopsy or a new biopsy obtained before the initiation of the treatment.
* Patients must have measurable disease other than the injection site or biopsy site.
* 18 years of age or older.
* Karnofsky Performance Status (KPS) of > 70.
* Adequate bone marrow function: WBC >2000/uL, platelet count >75,000/mm3; ANC>1000.
* Adequate hepatic function: bilirubin <= 1.5 mg/dL; SGOT/SGPT<2.5x upper limit of normal
* Adequate renal function: serum creatinine <= 2.0mg/dL.
* Required wash out periods for prior therapy:
* Topical therapy: 2 weeks
* Chemotherapy: 4 weeks (12 weeks for purine analogs)
* Radiotherapy (including photo therapy): 4 weeks
* Other systemic biological therapy: 4 weeks
* Other investigational therapy: 4 weeks
* Patients of reproductive potential and their partners must agree to use an effective (>90% reliability) form of contraception during the study and for 4 weeks following the last study drug administration.
* Women of reproductive potential must have negative urine pregnancy test.
* Life expectancy greater than 4 months.
* Able to comply with the treatment schedule.

Exclusion Criteria:

* Pre-existing autoimmune or antibody mediated disease including: systemic lupus, erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, etc, but excluding controlled thyroid disease, or the presence of autoantibodies without clinical autoimmune disease.
* Known history of human immunodeficiency virus (HIV) or hepatitis B or C.
* CNS metastases
* Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix.
* Current anticoagulant therapy (ASA<= 325 mg/day allowed).
* Significant cardiovascular disease (i.e., NYHA class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias).
* Pregnant or lactating.
* Prior therapy with allogeneic stem cell transplant.
* Any other medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility of intratumoral dendritic cell vaccination | 2 years

SECONDARY OUTCOMES:
Clinical activity-response in local and distant lesions | 2 years
Immunological response with conventional CTL assay, proliferation assay and microarray-based immune gene profiling using peripheral blood and/or biopsied tumor | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Palucka, MD, PhD, Study Director